CLINICAL TRIAL: NCT04069988
Title: Exploring the Effect of Baduanjin on the Metabolic Parameters and Body Mass Index of People With Schizophrenia: A Randomized Controlled Trial
Brief Title: Exploring the Effect of Baduanjin on the Metabolic Parameters and Body Mass Index of People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TSGHIRB2-105-05-005
Record Dates: First submitted 2019-08-25; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Randomized Controlled Trial
Keywords: Baduanjin; body mass index; metabolic parameters; metabolic syndrome; schizophrenia
MeSH Terms: conditions — Metabolic Syndrome; Schizophrenia

STUDY DESIGN:
Intervention Model Description: The participants were divided into experimental and control groups through block randomization.
Who Masked: Participant
Masking Description: The data of the five metabolic indexes, height, and bodyweight were collected by a research assistant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group (CG) received routine care and was required to physical activity for thirty minutes
- Baduanjin program (Experimental): The entire program continued for 6 months (March to October 2016), and the intervention was performed for 60 min 3 times for 12-weeks ; particular attention was paid to the disease characteristics of the patients with chronic schizophrenia and to preventing excessive fatigue. Every session began with a 20-min warm-up, followed by 20 min of Baduanjin program, and ended with a cool-down session. The participants were instructed, with the assistance of a video, to practice Baduanjin program in a group by two authors who are experienced in the psychiatric nurses and had been trained in this program.
  Interventions: Behavioral: Baduanjin program

INTERVENTIONS:
Behavioral: Baduanjin program — This exercise program aimed to increase patient participation and control their metabolic parameters and body mass index through Baduanjin program. The entire program continued for 6 months (March to October 2016), and the intervention was performed for 60 min 3 times for 12-weeks; particular attention was paid to the disease characteristics of the patients with chronic schizophrenia and to preventing excessive fatigue. Every session began with a 20-min warmup, followed by 20 min of Baduanjin program, and ended with a cool-down session. The participants were instructed, with the assistance of a video, to practice Baduanjin program in a group by two authors who are experienced in the psychiatric nurses and had been trained in this program.
  Arms: Baduanjin program

SUMMARY:
Baduanjin seems to be effective for improving body mass index and fasting sugar in male individuals with schizophrenia.

Aim This study was to explore the effect of Baduanjin on the five metabolic parameters and body mass index in participants with chronic schizophrenia.

Methods We recruited 92 participants from 3 chronic wards and nursing homes in eastern and northern Taiwan. Participants were assigned by blocked randomization into experimental group and control group. Those in the experimental group received 60 minutes, three times a week for 12 weeks of Baduanjin program training, while those in the control group received physical activity for thirty minutes. We collected the blood pressure, fasting blood sugar, triglyceride, high density cholesterol, waist circumference, and body mass index three times: before the intervention, end of the intervention immediately and 3-month follow up. Chi-squared and independent samples t test were used to compare the groups differences in the demographic characteristics and outcome indicators at the baseline for male and female separately. Demographic variables were controlled. Generalized Estimating Equations (GEE) were used to examine the effects of groups, time, group and time interaction by sex.

DETAILED DESCRIPTION:
This study explored the effect of Baduanjin on metabolic parameters and body mass index in people with schizophrenia. We recruited 92 participants from 3 rehabilitation units in Taiwan. Participants were assigned by blocked randomization into an experimental group or control group. Those in the experimental group received 60 minutes of Baduanjin three times a week for 12-weeks, while those in the control group received physical activity for thirty minutes. We assessed five metabolic parameters and body mass index at three timepoints: baseline, posttest and 3-month follow up.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of schizophrenia
2. between 20-65 years of age
3. BMI ≥ 24 kg/m2 or at least one metabolic parameter abnormality
4. ability to listen, speak and write Chinese
5. no additional exercise beyond normal exercise.

Exclusion Criteria:

1. patients in acute phase requiring hospitalization;
2. patients with severe and unstable

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
body Mass Index | 6 months
  BMI is defined as Body weight(kilograms) divided by height (meter) squared
Fasting blood sugar | 6 months
  Change from Baseline Fasting blood sugar (mg/dl) at 3 months and 6 months
Waist circumference | 6 months
  Change from Baseline Waist circumference (inches) at 3 months and 6 months
triglyceride | 6 months
  Change from Baseline triglyceride (mg/dl) at 3 months and 6 months
Blood pressure | 6 months
  Change from Baseline Blood pressure (mmHg) at 3 months and 6 months
high-density lipoprotein | 6 months
  Change from Baseline high-density lipoprotein (mg/dl) at 3 months and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan